CLINICAL TRIAL: NCT02442492
Title: STRIDER Canada: A Randomized Controlled Trial of Sildenafil Therapy In Dismal Prognosis Early-Onset Intrauterine Growth Restriction (Canada)
Brief Title: Sildenafil Therapy In Dismal Prognosis Early-Onset Intrauterine Growth Restriction
Acronym: STRIDERCan
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Trial terminated following Dutch DSMB recommendation for their Study
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kenneth Lim, Study Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H15-00899
Record Dates: First submitted 2015-05-05; First posted 2015-05-13 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Intrauterine Growth Restriction (IUGR); Fetal Growth Restriction (FGR)
Keywords: sildenafil; IUGR; FGR; STRIDER
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Active Comparator): Sildenafil 25 mg tablets three times daily orally from randomization until delivery or 31+6 weeks of gestational age, whichever is sooner.
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): Placebo 25 mg tablets three times daily orally from randomization until delivery or 31+6 weeks of gestational age, whichever is sooner.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil — Sildenafil 25 mg tablets three times daily orally from randomization until delivery or 31+6 weeks of gestational age, whichever is sooner.
  Arms: Sildenafil
Drug: Placebo — Placebo 25 mg tablets three times daily orally from randomization until delivery or 31+6 weeks of gestational age, whichever is sooner.
  Arms: Placebo

SUMMARY:
Early-onset placental intrauterine growth restriction (EO IUGR) is associated with a high risk of perinatal morbidity and mortality. In association with reduced circulating placental growth factor (PlGF) EO IUGR results from abnormal placentation with inadequate remodelling of the maternal uteroplacental arteries. There is no known treatment for placental IUGR. Management involves intensive fetal surveillance with delivery with evidence of serious fetal compromise. However, remote from term, delivery is associated with significant perinatal mortality and morbidity. Sildenafil vasodilates the uteroplacental vessels of IUGR-affected pregnancies and may represent a novel therapy.

DETAILED DESCRIPTION:
STRIDER Canada is one of a consortium of STRIDER randomised controlled trials (RCTs) each of which is designed to determine whether or not maternal treatment with oral sildenafil citrate improves perinatal outcomes in pregnancies complicated by EO IUGR without increasing risks to the mother.

STRIDER Canada is designed as investigator-initiated double-blind, randomised placebo-controlled trial of 90 women with a diagnosis of early-onset intrauterine growth restriction with an intention-to-treat analysis. 90 Women with affected pregnancies will be recruited and randomised to receive either sildenafil or placebo.

Women reviewed in the participating fetal medicine with a diagnosis of a pregnancy affected by early-onset IUGR between 18+0 and 27+6 weeks of gestation and serum PlGF levels less than 5th percentile for gestational age will be considered for randomisation. In Canadian STRIDER, the treatment with either sildenafil or placebo (25 mg 3 times per day) will be applied from the time of randomisation until delivery, or up to 31+6 weeks of gestation whichever comes first.

All patients randomly assigned to one of the treatments will be analysed together, regardless of whether or not they completed or received that treatment, on an intention to treat basis.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age from 18+0 - 27+6 weeks

AND

* EO IUGR, defined as

  1. ultrasound (U/S) measurement of the fetal abdominal circumference (AC) <10th percentile for gestational age and/or documented reduced fetal growth velocity complicating either a prior EO IUGR with adverse perinatal outcome or abnormal uterine artery waveform in the index pregnancy;

     OR
  2. U/S estimate of fetal weight (EFW) <700g

AND

* Serum PlGF < 5th percentile for gestational age

Exclusion Criteria:

* known fetal aneuploidy
* known fetal anomaly/syndrome/congenital infection confirmed at the time of enrolment
* decision made to terminate pregnancy
* current cocaine or vasoconstrictor use (e.g. crystal meth) (risk of acute cardiac events)
* contraindication to sildenafil therapy, e.g. known significant maternal cardiac disease, left ventricular outflow tract obstruction, concomitant treatment with nitrates or previous allergy to sildenafil
* known HIV positive status (due drug-drug interaction between sildenafil and antiretrovirals)
* receiving peripheral alpha-blockers (e.g. prazosin)
* prior participation in a STRIDER trials
* pre-eclampsia or gestational hypertension diagnosed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
compare the gestational age at delivery (d) between sildenafil- and placebo-treated groups | 6 weeks after postpartum

SECONDARY OUTCOMES:
live birth | at delivery if alive
survival to hospital discharge | measured at the final hospital discharge (average upto 6 weeks postpartum)
intact survival (defined as survival to estimated due date (EDD) without evidence of severe central nervous system [CNS] injury [by ultrasound and/or magnetic resonance imaging (MRI)]) | measured at estimated due date (EDD)
composite non-CNS (Central Nervous System) severe morbidity (one/more of bronchopulmonary dysplasia requiring supplemental oxygen on hospital discharge, ≥grade 3 retinopathy of prematurity, or necrotising enterocolitis) | up to 6 weeks after postpartum or final discharge which ever is sooner

OTHER OUTCOMES:
Maternal - symptomatic hypotension | up to 6 weeks after postpartum or final discharge which ever is sooner
Maternal - pre-eclampsia | from randomisation to delivery (expected to be assessed weekly)
Maternal - mode of delivery | At delivery
Maternal - haemorrhage requiring transfusion | At delivery
Maternal - maternal plasma PlGF. | from randomisation to delivery (expected to be assessed weekly)
Maternal - uterine artery Doppler indices | from randomisation to delivery (expected to be done weekly)
Perinatal - fetal growth velocity | from randomisation to delivery (expected to be done weekly)
Perinatal - fetal Doppler | from randomisation to delivery (expected to be done weekly)
Perinatal - amniotic fluid | At randomisation, if done
Perinatal - fetal heart indices | rom randomisation to delivery (expected to be done weekly)

CONTACTS AND LOCATIONS:
Overall Officials: Peter von Dadelszen, BMedSc, MBChB, DipObst, DPhil,, Principal Investigator — University of British Columbia; Kenneth Lim, MD FRCSC, Principal Investigator — University of British Columbia
Locations (5):
- Canada (5):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - BC Women's Hospital/University of British Columbia, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - CHU de Quebec - Universite Laval, Québec, Quebec

REFERENCES:
- [Derived] von Dadelszen P, Audibert F, Bujold E, Bone JN, Sandhu A, Li J, Kariya C, Chung Y, Lee T, Au K, Skoll MA, Vidler M, Magee LA, Piedboeuf B, Baker PN, Lalji S, Lim KI. Halting the Canadian STRIDER randomised controlled trial of sildenafil for severe, early-onset fetal growth restriction: ethical, methodological, and pragmatic considerations. BMC Res Notes. 2022 Jul 7;15(1):244. doi: 10.1186/s13104-022-06107-y. PMID 35799272
- [Derived] Pels A, Kenny LC, Alfirevic Z, Baker PN, von Dadelszen P, Gluud C, Kariya CT, Mol BW, Papageorghiou AT, van Wassenaer-Leemhuis AG, Ganzevoort W, Groom KM; international STRIDER Consortium. STRIDER (Sildenafil TheRapy in dismal prognosis early onset fetal growth restriction): an international consortium of randomised placebo-controlled trials. BMC Pregnancy Childbirth. 2017 Dec 28;17(1):440. doi: 10.1186/s12884-017-1594-z. PMID 29282009